CLINICAL TRIAL: NCT04252365
Title: A Randomized Controlled, Phase II Trial Comparing Sintilimab and Pembrolizumab at First-line Setting in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Sintilimab Versus Pembrolizumab for Advanced-stage Non-Small-Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1901
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Nsclc
Keywords: PD-1 inhibitors, immunotherapy, NSCLC, PD-L!
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm 1 (Experimental): Patients with PD-L1 high expression (TPS≥50%) receive Sintilimab injection 200mg i.v. on day 1 every three weeks (Q3W). Courses repeat every 21days in the absence of disease progression or unacceptable toxicity.
  Patients with PD-L1 low or negative expression (TPS<50%) receive Sintilimab injection 200mg i.v. in combination with platinum-based chemotherapy every three weeks (Q3W) for 4 cycles. After that, patients receive Sintilimab injection on day 1 Q3W during the maintenance phase (Cycle 5 onward). Courses repeat every 21days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Sintilimab
- arm 2 (Active Comparator): Patients with PD-L1 high expression (TPS≥50%) receive Pembrolizumab injection 200mg i.v. on day 1once every three weeks (Q3W). Courses repeat every 21days in the absence of disease progression or unacceptable toxicity.
  Patients with PD-L1 low or negative expression (TPS<50%) receive Pembrolizumab injection 200mg i.v. in combination with platinum-based chemotherapy every three weeks (Q3W) for 4 cycles. After that, patients receive Pembrolizumab injection on day 1 Q3W during the maintenance phase (Cycle 5 onward). Courses repeat every 21days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Sintilimab — Given i.v.
  Other Names: IBI308
  Arms: arm 1
Drug: Pembrolizumab — Given i.v.
  Other Names: Keytruda
  Arms: arm 2

SUMMARY:
This study is a single-center, randomized controlled, phase II clinical trial, aiming at giving a comparison of Sintilimab and Pembrolizumab in stage IIIB-IV NSCLC patients at first-line treatment setting.

DETAILED DESCRIPTION:
This trial has been set up with two arms. Screened patients would be included into one of the arms based on tumor PD-L1 expression. The purpose of this study is to compare the efficacy of the approved checkpoint inhibitor pembrolizumab and home-made drug Sintilimab in patients with advanced NSCLC whose tumor have high PD-L1 expression and low or negative expression.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years. Signed Informed Consent Form.
2. Stage IV NSCLC confirmed by histology/ cytology or Stage IIIB-IIIC NSCLC that could not be treated with radical radiation therapy (8th edition of IASLC Lung Cancer Staging System).
3. Fresh tumor tissue or paraffin tissue within 6 months is adequate for PD-L1 expression (TPS) testing in the central laboratory.
4. Tumor tissue without EGFR mutation or ALK rearrangement must be confirmed.
5. Per RECIST 1.1 the efficacy evaluation criteria for solid tumors, at least one radiologically measurable lesion which was not treated with radiotherapy or had obvious disease progression after radiotherapy.
6. Patients who received no systemic chemotherapy or any other systemic treatment for advanced NSCLC. For patients who received preoperative neoadjuvant chemotherapy or postoperative adjuvant chemotherapy or radical chemoradiotherapy, if the disease progresses occurred one six months after the last treatment, they can be enrolled. Patients who received targeted therapy or immunotherapy can not be enrolled.

Exclusion Criteria:

1. Active hepatitis B. Active hepatitis B is defined as HBsAg positive and the detected HBV-DNA copy number is larger than the upper limit of normal value in the laboratory of the study site.
2. Currently or prior clinically active interstitial lung disease. Currently active pneumonia. Current radiation pneumonitis for which corticosteroid treatment is required.
3. Known HIV antibody positive, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation.
4. Fever and the body temperature is above 38°C or clinically significant infection within 1 week prior to the enrollment.
5. Active tuberculosis. Evidence of severe or uncontrollable systemic diseases (such as severe mental, neurological diseases, seizure, or dementia, unstable or non-compensatory respiratory, cardiovascular, hepatic or renal diseases, and uncontrolled hypertension [CTCAE Grade 2 hypertension or above after drug treatment]).
6. Patients with active bleeding or new thrombotic diseases who are orally taking with anticoagulant drugs or have bleeding tendency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years
  Defined as the percentage of patients whose tumors have a complete or partial response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long Wu, Study Chair — Guangdong Association of Clinical Trials, GACT